CLINICAL TRIAL: NCT05572164
Title: Comparison On Efficiency Of Surgical Pleth Index-Guided Traditional Epidural And Dural Puncture Epidural Analgesia Techniques In Percutaneous Nephrolithotomy: A Randomised Double Blind Study
Brief Title: Comparison Of Epidural Analgesia Techniques In Percutaneous Nephrolithotomy With Surgical Pleth Index
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Clinical Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/576
Record Dates: First submitted 2022-09-13; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRADITIONAL EPIDURAL (Active Comparator): standard epidural technique used for intraoperative analgesia (the EPL group; local anesthetics will be delivered via epidural catheter guided by SPI to provide intraoperative analgesia
  Interventions: Procedure: TRADITIONAL EPIDURAL
- DURAL PUNCTURE EPIDURAL (Active Comparator): group on whom dural puncture epidural technique used for intraoperative analgesia ( the DPL group; local anesthetics will be delivered via an epidural catheter placed after a dural pucture performed with the SPI guidance to provide intraoperative analgesia)
  Interventions: Procedure: DURAL PUNCTURE EPIDURAL

INTERVENTIONS:
Procedure: TRADITIONAL EPIDURAL — epidural technique used for intraoperative analgesia (the EPL group; local anesthetics will be delivered via epidural catheter guided by SPI to provide intraoperative analgesia)
  Arms: TRADITIONAL EPIDURAL
Procedure: DURAL PUNCTURE EPIDURAL — group on whom dural puncture epidural technique used for intraoperative analgesia ( the DPL group; local anesthetics will be delivered via an epidural catheter placed after a dural pucture performed with the SPI guidance to provide intraoperative analgesia)
  Arms: DURAL PUNCTURE EPIDURAL

SUMMARY:
Primary aim of this study is to evaluate affect of SPI guided antinociception on total intraoperative consumption of local aneshesics during analgesia. Secondary aims are defining time interval between LA administration and SPI value dropping under 50 and hemodynamy. Tertiary results are total mean local anesthesic consumption per hour, mean LA bolus number, total norepinephrine, ephedrine and atrophine consumption, mean intraoperative heart rate, mean arterial pressure, BIS and minimal alveolar concentration, percentage of intraoperative surgery time during which SPI>50, time passed until first post operative analgesia need, time needed to be discharged from PACU after operation (evaluated via Aldrte score) and post operative side effects (nausea, vomiting, sedatition and piruritis)

ELIGIBILITY:
Inclusion Criteria:

* aged 18-60
* ASA I-III
* grade I unilateral PNL

Exclusion Criteria:

* BMI > 40 kg/m2
* drug or alcohol abuse history in the last 6 mounts
* chronic opoid usage or had chronic pain longer than 6 weeks
* peripheral and central neurological disorders
* preoperative hemodynamic disorders
* irregular sinus rhythm and pace makers
* diabetes, severe lung and major liver diseases with increasing biluribin
* use of anti-muscarinics, α2-adrenergic agonists, β1-adrenergic agonists, anti arrhythmic; who used chronic psychoactive drugs in last 90 days
* who are pregnant and breast feeding
* not willing to participate
* allergic or intolerant to any of the drugs in the study
* procedures that take less than 2 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
consumption of local aneshesics | intraoperative
  to evaluate affect of SPI guided antinociception on total intraoperative consumption of local aneshesics during analgesia

SECONDARY OUTCOMES:
time interval and SPI value dropping | intraoperative
  defining time interval between LA administration and SPI value dropping under 50 and hemodynamy
local anesthesic consumption | during the procedure/surgery and during 30 minutes of PACU stay
  total mean local anesthesic consumption per hour, mean LA bolus number, total norepinephrine, ephedrine and atrophine consumption, mean intraoperative heart rate, mean arterial pressure, BIS and minimal alveolar concentration, percentage of intraoperative surgery time during which SPI>50, time passed until first post operative analgesia need, time needed to be discharged from PACU after operation (evaluated via Aldrte score) and post operative side effects (nausea, vomiting, sedatition and piruritis)

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Dostbil, Study Director — Ataturk University